CLINICAL TRIAL: NCT02616120
Title: Efficacy and Safety of SQJZ Herbal Mixtures on Non-motor Symptoms in Parkinson's Disease Patients
Brief Title: Effect of SQJZ Herbal Mixtures on Non-motor Symptoms of Parkinson's Disease
Acronym: ESNMS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Jinzhou Tian, vice-president, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECPJ-BDY-2014-27; SHOUFA 2014-1-4 (Other: Beijing Municipal Commission of Health and Family Planning)
Record Dates: First submitted 2015-11-20; First posted 2015-11-26 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Parkinson's Disease
Keywords: Herbal therapy; Parkinson's Disease; Non-motor Symptoms; Randomized controlled trial
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): placebo identified to SQJZ herbal mixtures, 29.375g, 2 times per day.for 12 weeks.
  Interventions: Drug: Placebo
- SQJZ herbal mixtures (Active Comparator): SQJZ herbal mixtures 29.375g, 2 times per day.for 12 weeks.
  Interventions: Drug: SQJZ herbal mixtures

INTERVENTIONS:
Drug: SQJZ herbal mixtures — The SQJZ herbal mixtures is Chinese herb extracts. It contains Rehmannia glutinosa Libosch，Astragalus membranaceus (Fisch.) Bunge etc.( 29.375g, 2 times per day)
  Arms: SQJZ herbal mixtures
Drug: Placebo — placebo contains 5%SQJZ herbal mixtures and 95% dextrin,identified to SQJZ herbal formula (29.375g, 2 times per day)
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the efficacy and safety of SQJZ Herbal Mixtures on non-motor symptoms of PD patients.

DETAILED DESCRIPTION:
This will be a multicentre, double-blind, placebo-controlled, parallel-group trial. Patients will be randomly assigned via an random number table to either the SQJZ herbal mixtures or placebo in a 2:1 ratio. Randomization will be stratify by age and gender. All participants are asked to maintain the regular medication schedule during the 12-week intervention. Assessments are conducted prior to the intervention and at 4-week, 8-week and 12-week directly after the intervention. Also, long-term effects will be assessed at 24 weeks of follow-up (from post-enrolment). The assessments will be performed by a blinded investigator who is not involved in the randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has idiopathic Parkinson's disease with diagnostic standard of (UKPDC)
2. Subject has a Hoehn and Yahr stage score ≤4
3. Subject is male or female, ≥18 years of age，and≤80 years.
4. Subject has a total Non-Motor Symptoms Scale (NMSS) score ≥40
5. If the subject is receiving levodopa (L-DOPA),anticholinergics, monoamine oxidase (MAO) B inhibitors, or amantadine, he/she must have been on a stable dose for at least 28 days prior to the Baseline Visit and must be maintained on that dose for the duration of the study
6. Subject agree to sign an informed consent.

Exclusion Criteria:

1. Subject is receiving therapy with anti-Parkinson's disease drugs(include levodopa (L-DOPA), amantadine, anticholinergics, monoamine oxidase (MAO) B inhibitors, dopamine receptor agonists or catechol-O-methyltransferase inhibitor),which is not under the guidance of professional doctors,either concurrently or within 28 days prior to the Baseline Visit.
2. Subject is receiving therapy with 1 of the following drugs, either concurrently or within 28 days prior to the Baseline Visit: alpha-methyl dopa, metoclopramide, reserpine, sibelium ,neuroleptics (except specific atypical neuroleptics: olanzapine, ziprasidone, aripiprazole, clozapine, and quetiapine), monoamine oxidase-A (MAO-A) inhibitors, methylphenidate, amphetamine.
3. Subject is receiving central nervous system (CNS) therapy (eg, sedatives, hypnotics, selective serotonin reuptake inhibitors [SSRIs], anxiolytics, or other sleep-modifying medication) unless dose has been stable daily for at least 28 days prior to the Baseline Visit and is likely to remain stable for the duration of the study
4. Subject has visual hallucination,and the visual hallucination happened within 1 year after been diagnosed with PD.
5. Subject has delirium。
6. Subject has Other digestive, Urological , blood system , endocrine , immune system or cardiopulmonary problems that in the view of the researchers.
7. Subject has Serum creatinine≥97umol/L；or the alanine aminotransferase(ALT) ≥40U/L;or aspartate aminotransferase≥40U/L。
8. Subject has a epilepsy history.
9. Subject has evidence of an impulse control disorder, a history of mental illness, thoughts or behaviors of suicide.
10. According to the assessment of the investigator,Subject cann't complete the study due to poor compliance, drug or Alcohol abuse.
11. Subject is participating in other clinical trials or Participated in the past 2 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
changes of The Nonmotor Symptoms Scale (NMSS) from baseline after 12-weeks treatment. | baseline, 4-week, 8-week, 12-week and 24-week.
  The Nonmotor Symptoms Scale (NMSS) is a validated tool for rating frequency and severity of nonmotor symptoms in Parkinson's Disease (PD). The severity and frequency of the subject's nonmotor symptoms is assessed by the investigator in the following 9 domain categories: cardiovascular, including falls; sleep/fatigue; mood/cognition; perceptual problems/hallucinations; attention/memory; gastrointestinal tract; urinary; sexual function; miscellaneous. Severity and frequency are rated using a 4-point scale ranging from 0 (none) to 3 (severe; major source of distress or disturbance to subject) for severity and from 1 (rarely) to 4 (very frequent [daily or all the time]) for frequency. The total NMSS score ranges from 0 to 350. A negative change from Baseline to end of Maintenance indicates an improvement in NMSS. The NMSS was assessed at introduction period, baseline, 4-week, 8-week, 12-week and 24-week.

SECONDARY OUTCOMES:
changes of The Unified Parkinson's Disease Rating Scale (UPDRS) from baseline after 12-weeks treatment. | baseline, 4-week, 8-week, 12-week and 24-week.
  This questionnaire is a scale for the assessment of function in Parkinson's Disease.It is derived from Part I (Mentation, Behavior and Mood), Part II (Activities of Daily Living) and Part III (Motor Examination). Part I assesses 4 functions; Part II assesses 13 activities of daily living; Part III assesses 14 motor symptoms. Each item is rated on a scale from 0 (normal) to 4 (severe). The minimum total score possible is 0 and the maximum total score possible is 176. Each subject was independently rated by two observers at each study visit and a mean score was calculated for analysis.
changes of The Parkinson's Disease Questionnaire-39 (PDQ-39) from baseline after 12-weeks treatment. | baseline, 12-week and 24-week
  This questionnaire is a measure of quality of life adapted for people with PD . It consists of 39 statements that cover eight domains associated with health, such as mobility and emotionality, that can be influenced by PD. Patients can reply by ticking the relevant answer that indicates whether they experienced problems during the past month (five boxes from 'never' to 'always').

CONTACTS AND LOCATIONS:
Overall Officials: JinZhou Tian, MD,PhD, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen hospital, Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China